CLINICAL TRIAL: NCT01691898
Title: A Randomized, Open-Label, Multicenter, Phase II Trial Evaluating the Safety and Activity of Pinatuzumab Vedotin (DCDT2980S) in Combination With Rituximab or Polatuzumab Vedotin (DCDS4501A) in Combination With Rituximab and a Non-Randomized Phase Ib/II Evaluation of Polatuzumab Vedotin in Combination With Obinutuzumab in Patients With Relapsed or Refractory B-Cell Non-Hodgkin's Lymphoma
Brief Title: A Study of Pinatuzumab Vedotin (DCDT2980S) Combined With Rituximab or Polatuzumab Vedotin (DCDS4501A) Combined With Rituximab or Obinutuzumab in Participants With Relapsed or Refractory B-Cell Non-Hodgkin's Lymphoma (NHL)
Acronym: ROMULUS
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO27834; 2011-004377-84 (EudraCT Number)
Record Dates: First submitted 2012-09-16; First posted 2012-09-25 (Estimated); Results first posted 2018-04-19 (Actual); Last update posted 2020-02-21 (Actual); Status verified 2020-02

CONDITIONS: Follicular Lymphoma; Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse | interventions — obinutuzumab; pinatuzumab vedotin; polatuzumab vedotin; Rituximab

ARMS (6):
- Arm A (FL+DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab (Experimental): For the first 2 cycles, RTX 375 milligrams per square meter (mg/m^2) will be given by intravenous (IV) infusion on Day 1 and pinatuzumab vedotin 2.4 milligrams per kilogram (mg/kg) will be administered by IV infusion on Day 2 to Arm A participants (with r/r FL and DLBCL). In the absence of any infusion-related adverse events, RTX and pinatuzumab may be administered on the same day (Day 1) in subsequent cycles beginning with the third cycle. Participants who develop disease progression (PD) will be further treated with RTX 375 mg/m^2 followed by polatuzumab vedotin 2.4 mg/kg IV infusion on Day 1, beginning no later than 42 days after the last dose of the prior study treatment until a second PD event relative to the tumor assessment, documenting PD on the initial study treatment, clinical deterioration, and/or intolerance to the crossover treatment for up to a maximum of 1 year (17 cycles on an every-21-day schedule).
  Interventions: Drug: Pinatuzumab Vedotin; Drug: Polatuzumab Vedotin; Drug: Rituximab
- Arm B (FL+DLBCL): RTX+Polatuzumab,Then RTX+Pinatuzumab (Experimental): For the first 2 cycles, RTX 375 mg/m^2 will be given by IV infusion on Day 1 and polatuzumab vedotin 2.4 mg/kg will be administered by IV infusion on Day 2 to Arm B participants (with r/r FL and DLBCL). In the absence of any infusion-related adverse events, RTX and polatuzumab may be administered on the same day (Day 1) in subsequent cycles beginning with the third cycle. Participants who develop PD would be further treated with RTX 375 mg/m^2 followed by pinatuzumab vedotin 2.4 mg/kg IV infusion on Day 1, beginning no later than 42 days after the last dose of the prior study treatment until a second PD event relative to the tumor assessment, documenting PD on the initial study treatment, clinical deterioration, and/or intolerance to the crossover treatment for up to a maximum of 1 year (17 cycles on an every-21-day schedule).
  Interventions: Drug: Pinatuzumab Vedotin; Drug: Polatuzumab Vedotin; Drug: Rituximab
- Cohort C (FL): RTX + Polatuzumab (Experimental): For the first 2 cycles, RTX 375 mg/m^2 will be given by IV infusion on Day 1 and polatuzumab vedotin 1.8 mg/kg will be administered by IV infusion on Day 2 to Cohort C participants (with r/r FL). In the absence of any infusion-related adverse events, RTX and polatuzumab may be administered on the same day (Day 1) in subsequent cycles beginning with the third cycle for up to a maximum of 1 year (17 cycles on an every-21-day schedule) or significant toxicity, PD, or withdrawal from study.
  Interventions: Drug: Polatuzumab Vedotin; Drug: Rituximab
- Cohort E (FL+DLBCL): Obinutuzumab + Polatuzumab (Experimental): For the first cycle, obinutuzumab will be given by IV infusion on Days 1, 8, and 15. Polatuzumab vedotin 1.8 mg/kg IV infusion will be given on Day 2 of the first cycle to Cohort E participants (with r/r FL and DLBCL). In the absence of any infusion-related adverse events, obinutuzumab and polatuzumab vedotin may be administered on the same day (Day 1) in subsequent cycles beginning with the second cycle up to a maximum of 8 cycles or significant toxicity, PD, or withdrawal from study.
  Interventions: Drug: Obinutuzumab; Drug: Polatuzumab Vedotin
- Cohort G (Expansion, FL): Obinutuzumab + Polatuzumab (Experimental): For the first cycle, obinutuzumab will be given by IV infusion on Days 1, 8, and 15. Polatuzumab vedotin 1.8 mg/kg IV infusion will be given on Day 2 of the first cycle to Cohort G participants (with r/r FL). In the absence of any infusion-related adverse events, obinutuzumab and polatuzumab vedotin may be administered on the same day (Day 1) in subsequent cycles beginning with the second cycle of the dose-expansion period to cohort G participants up to a maximum of 8 cycles or significant toxicity, PD, or withdrawal from study.
  Interventions: Drug: Obinutuzumab; Drug: Polatuzumab Vedotin
- Cohort H (Expansion, DLBCL): Obinutuzumab + Polatuzumab (Experimental): For the first cycle, obinutuzumab will be given by IV infusion on Days 1, 8, and 15. Polatuzumab vedotin 1.8 mg/kg IV infusion will be given on Day 2 of the first cycle to Cohort H participants (with r/r DLBCL). In the absence of any infusion-related adverse events, obinutuzumab and polatuzumab vedotin may be administered on the same day (Day 1) in subsequent cycles beginning with the second cycle of the dose-expansion period to cohort H participants up to a maximum of 8 cycles or significant toxicity, PD, or withdrawal from study.
  Interventions: Drug: Obinutuzumab; Drug: Polatuzumab Vedotin

INTERVENTIONS:
Drug: Obinutuzumab — Obinutuzumab 1000 mg will be administered by IV infusion on Days 1, 8, 15 of first 21-Day cycle and on Day 1 of subsequent 21-day cycles for up to 8 cycles.
  Other Names: GA101, Gazyva, Gazyvaro
  Arms: Cohort E (FL+DLBCL): Obinutuzumab + Polatuzumab; Cohort G (Expansion, FL): Obinutuzumab + Polatuzumab; Cohort H (Expansion, DLBCL): Obinutuzumab + Polatuzumab
Drug: Pinatuzumab Vedotin — Pinatuzumab Vedotin 1.8 or 2.4 mg/kg administered by IV infusion on Day 1 or 2 of every 21-day cycle.
  Other Names: DCDT2980S
  Arms: Arm A (FL+DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab; Arm B (FL+DLBCL): RTX+Polatuzumab,Then RTX+Pinatuzumab
Drug: Polatuzumab Vedotin — Polatuzumab Vedotin 1.8 or 2.4 mg/kg administered by IV infusion on Day 1 or 2 of every 21-day cycle.
  Other Names: DCDS4501A
Drug: Rituximab — RTX 375 mg/m^2 administered by IV infusion on Day 1 of every 21-day cycle.
  Other Names: MabThera/Rituxan
  Arms: Arm A (FL+DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab; Arm B (FL+DLBCL): RTX+Polatuzumab,Then RTX+Pinatuzumab; Cohort C (FL): RTX + Polatuzumab

SUMMARY:
This multicenter, open-label study will evaluate the safety and efficacy of pinatuzumab vedotin (DCDT2980S) or polatuzumab vedotin (DCDS4501A) in combination with rituximab (RTX), as well as of polatuzumab vedotin in combination with obinutuzumab in participants with relapsed or refractory (r/r) follicular lymphoma (FL) and r/r diffuse large B-cell lymphoma (DLBCL).

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2
* Life expectancy of at least 12 weeks
* History of histologically documented r/r Grades 1 to 3a FL, or r/r DLBCL
* Availability of an archival or freshly biopsied tumor tissue sample must be confirmed for study enrollment
* Have a clinical indication for treatment as determined by the investigator
* Must have at least one bi-dimensionally measurable lesion (greater than [>] 1.5 centimeters [cm] in its largest dimension by CT scan or Magnetic Resonance Imaging [MRI])

Exclusion Criteria:

* Prior use of any monoclonal antibody, radio-immuno-conjugate or antibody drug conjugate within 4 weeks before study start
* Treatment with radiotherapy, chemotherapy, immunotherapy, immunosuppressive therapy, or any investigational anti-cancer agent within 2 weeks prior study start
* Adverse events except for sensory neuropathy from any previous treatments must be resolved or stabilized to Grade less than equal to (</=) 2 prior study start
* Completion of autologous stem cell transplant (SCT) within 100 days prior study start
* Prior allogeneic SCT
* Eligibility for autologous SCT (participants with r/r DLBCL)
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy (or recombinant antibody-related fusion proteins)
* History of other malignancy that could affect compliance with the protocol or interpretation of results
* Current or past history of central nervous system lymphoma
* Current Grade >1 peripheral neuropathy
* Vaccination with a live vaccine within 28 days prior to treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2012-09-27 (Actual); Primary Completion 2017-03-08 (Actual); Study Completion 2019-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (41):
- United States (26):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Stanford Cancer Center, Stanford, California
  - Colorado Blood Cancer Institute (CBCI) at Presbyterian/ St. Luke's Medical Center, Denver, Colorado
  - Georgetown University Medical Center Lombardi Cancer Center, Washington D.C., District of Columbia
  - Florida Cancer Specialists - Fort Myers (Colonial Center Dr), Fort Myers, Florida
  - Florida Cancer Specialists; Sarasota, Sarasota, Florida
  - Univ of Michigan Med School; Hematology Oncology, Ann Arbor, Michigan
  - Comprehensive Cancer Centers of Nevada - Eastern Avenue, Las Vegas, Nevada
  - Hematology Oncology Associates; Carol G. Simon Ctr, Morristown, New Jersey
  - Regional Cancer Care Associates LLC - Morristown, Morristown, New Jersey
  - Roswell Park Cancer Inst., Buffalo, New York
  - New York University Cancer Cen, New York, New York
  - Oncology Hematology Care Inc, Cincinnati, Ohio
  - Willamette Valley Cancer Ctr - 520 Country Club, Eugene, Oregon
  - Oregon Health Sciences Uni, Portland, Oregon
  - Sarah Cannon Cancer Center - Tennessee Oncology, Pllc, Nashville, Tennessee
  - Texas Oncology-Baylor Sammons Cancer Center, Dallas, Texas
  - Cancer Care Centers of South Texas, San Antonio, Texas
  - Texas Transplant Inst., San Antonio, Texas
  - Texas Oncology, P.A. - Tyler; Tyler Cancer Center, Tyler, Texas
  - Fairfax N Virginia Hem/Onc PC, Fairfax, Virginia
  - Oncology & Hematolgy Associates of SW Va Inc. - Roanoke, Roanoke, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Northwest Cancer Specialists - Vancouver, Vancouver, Washington
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington
  - Univ of Wisconsin-Madison, Madison, Wisconsin
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - McGill University; Sir Mortimer B Davis Jewish General Hospital; Oncology, Montreal, Quebec
- France (5):
  - Hopital Claude Huriez - CHU Lille, Lille
  - CHU Montpellier - Saint ELOI, Montpellier
  - Hopital Saint Louis ; Service d Oncologie Medicale Fougere 6 (Pr Misset), Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Henri Becquerel; Hematologie, Rouen
- Germany (3):
  - Uniklinik Heidelberg, Medizinische Klinik & Poliklinik V, Heidelberg
  - Universitätsmedizin Johannes Gutenberg Universität; Klinik u. Poliklinik f. Neurologie, Mainz
  - Klinikum d.Universität München Campus Großhadern, München
- Italy (3):
  - A.O. Universitaria Policlinico S.Orsola-Malpighi Di Bologna, Bologna, Emilia-Romagna
  - Irccs Istituto Nazionale Dei Tumori (Int);S.C. Medicina Oncologica 2, Milan, Lombardy
  - Azienda Ospedale San Giovanni, Turin, Piedmont
- Academisch Medisch Centrum; Hematologie, Amsterdam, Netherlands

REFERENCES:
- [Derived] Shi R, Lu T, Ku G, Ding H, Saito T, Gibiansky L, Agarwal P, Li X, Jin JY, Girish S, Miles D, Li C, Lu D. Asian race and origin have no clinically meaningful effects on polatuzumab vedotin pharmacokinetics in patients with relapsed/refractory B-cell non-Hodgkin lymphoma. Cancer Chemother Pharmacol. 2020 Sep;86(3):347-359. doi: 10.1007/s00280-020-04119-8. Epub 2020 Aug 8. PMID 32770353
- [Derived] Lu T, Gibiansky L, Li X, Li C, Shi R, Agarwal P, Hirata J, Miles D, Chanu P, Girish S, Jin JY, Lu D. Exposure-safety and exposure-efficacy analyses of polatuzumab vedotin in patients with relapsed or refractory diffuse large B-cell lymphoma. Leuk Lymphoma. 2020 Dec;61(12):2905-2914. doi: 10.1080/10428194.2020.1795154. Epub 2020 Jul 24. PMID 32705923
- [Derived] Morschhauser F, Flinn IW, Advani R, Sehn LH, Diefenbach C, Kolibaba K, Press OW, Salles G, Tilly H, Chen AI, Assouline S, Cheson BD, Dreyling M, Hagenbeek A, Zinzani PL, Jones S, Cheng J, Lu D, Penuel E, Hirata J, Wenger M, Chu YW, Sharman J. Polatuzumab vedotin or pinatuzumab vedotin plus rituximab in patients with relapsed or refractory non-Hodgkin lymphoma: final results from a phase 2 randomised study (ROMULUS). Lancet Haematol. 2019 May;6(5):e254-e265. doi: 10.1016/S2352-3026(19)30026-2. Epub 2019 Mar 29. PMID 30935953

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 289 participants were screened, out of which, 231 participants were enrolled into the study.
Groups:
- Arm A (FL+DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab: Participants with relapsed or refractory (r/r) follicular lymphoma (FL) and diffuse large B-cell lymphoma (DLBCL) received rituximab (RTX) at a dose of 375 milligrams per square meter (mg/m^2) administered via intravenous (IV) infusion on Day 1 and pinatuzumab vedotin at a dose of 2.4 milligrams per kilogram (mg/kg) administered via IV infusion on Day 2 for the first 2 cycles. RTX and pinatuzumab were administered on the same day (Day 1) in subsequent cycles beginning with the third cycle, in the absence of any infusion-related adverse events. Participants who developed disease progression (PD) were treated with RTX at 375 mg/m^2 and polatuzumab vedotin at 2.4 mg/kg via IV infusion on Day 1, beginning no later than 42 days after the last dose of the prior study treatment until a second PD event, clinical deterioration, and/or intolerance to the crossover treatment for up to a maximum of 1 year (maximum 17 cycles on an every-21-day schedule).
- Arm B (FL+DLBCL): RTX+Polatuzumab,Then RTX+Pinatuzumab: Participants with r/r FL and DLBCL received RTX at a dose of 375 mg/m^2 administered via IV infusion on Day 1 and polatuzumab vedotin at a dose of 2.4 mg/kg administered via IV infusion on Day 2 for the first 2 cycles. RTX and polatuzumab were administered on the same day (Day 1) in subsequent cycles beginning with the third cycle, in the absence of any infusion-related adverse events. Participants who developed PD were treated with RTX at 375 mg/m^2 and pinatuzumab vedotin at 2.4 mg/kg via IV infusion on Day 1, beginning no later than 42 days after the last dose of the prior study treatment until a second PD event, clinical deterioration, and/or intolerance to the crossover treatment for up to a maximum of 1 year (maximum 17 cycles on an every-21-day schedule).
- Cohort C (FL): RTX + Polatuzumab: Participants with r/r FL received RTX at a dose of 375 mg/m^2 administered via IV infusion on Day 1 and polatuzumab vedotin at a dose of 1.8 mg/kg administered via IV infusion on Day 2 for the first 2 cycles. In the absence of any infusion-related adverse events, RTX and polatuzumab were administered on the same day (Day 1) in subsequent cycles beginning with the third cycle for up to a maximum of 1 year (17 cycles on an every-21-day schedule) or significant toxicity, disease progression, or withdrawal from study.
- Cohort E (FL+DLBCL): Obinutuzumab + Polatuzumab: Participants with r/r FL and DLBCL received obinutuzumab at a dose of 1000 mg via IV infusion on Days 1, 8, 15 and polatuzumab vedotin at a dose of 1.8 mg/kg administered via IV infusion on Day 2 for the first cycle. In the absence of any infusion-related adverse events, obinutuzumab and polatuzumab vedotin were administered on the same day (Day 1) in subsequent cycles beginning with the second cycle for up to a maximum of 8 cycles or significant toxicity, disease progression, or withdrawal from study.
- Cohort G (Expansion, FL): Obinutuzumab + Polatuzumab: Participants with r/r FL received obinutuzumab at a dose of 1000 mg via IV infusion on Days 1, 8, 15 and polatuzumab vedotin at a dose of 1.8 mg/kg administered via IV infusion on Day 2 for the first cycle. In the absence of any infusion-related adverse events, obinutuzumab and polatuzumab vedotin were administered on the same day (Day 1) in subsequent cycles beginning with the second cycle for up to a maximum of 8 cycles or significant toxicity, disease progression, or withdrawal from study.
- Cohort H (Expansion, DLBCL): Obinutuzumab + Polatuzumab: Participants with r/r DLBCL received obinutuzumab at a dose of 1000 mg via IV infusion on Days 1, 8, 15 and polatuzumab vedotin at a dose of 1.8 mg/kg administered via IV infusion on Day 2 for the first cycle. In the absence of any infusion-related adverse events, obinutuzumab and polatuzumab vedotin were administered on the same day (Day 1) in subsequent cycles beginning with the second cycle for up to a maximum of 8 cycles or significant toxicity, disease progression, or withdrawal from study.
Period: Overall Study
Arm/Group | Arm A (FL+DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm B (FL+DLBCL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Cohort C (FL): RTX + Polatuzumab | Cohort E (FL+DLBCL): Obinutuzumab + Polatuzumab | Cohort G (Expansion, FL): Obinutuzumab + Polatuzumab | Cohort H (Expansion, DLBCL): Obinutuzumab + Polatuzumab
Started | 63 | 59 | 20 | 9 | 40 | 40
Completed | 16 | 15 | 11 | 4 | 26 | 5
Not Completed | 47 | 44 | 9 | 5 | 14 | 35
Not completed — Death | 34 | 32 | 6 | 3 | 8 | 31
Not completed — Adverse Event | 0 | 1 | 0 | 1 | 1 | 0
Not completed — Progression of Disease | 1 | 2 | 1 | 0 | 0 | 1
Not completed — Lost to Follow-up | 3 | 1 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 9 | 8 | 2 | 1 | 3 | 3
Not completed — Non-Compliance | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on safety-evaluable population, which included all participants who received at least 1 dose of all study treatment.
Groups:
- Arm A (FL+DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab: Participants with relapsed or refractory [r/r] FL and DLBCL received rituximab (RTX) at a dose of 375 milligrams per square meter (mg/m^2) administered via intravenous (IV) infusion on Day 1 and pinatuzumab vedotin at a dose of 2.4 milligrams per kilogram (mg/kg) administered via IV infusion on Day 2 for the first 2 cycles. RTX and pinatuzumab were administered on the same day (Day 1) in subsequent cycles beginning with the third cycle, in the absence of any infusion-related adverse events. Participants who developed disease progression (PD) were treated with RTX at 375 mg/m^2 and polatuzumab vedotin at 2.4 mg/kg via IV infusion on Day 1, beginning no later than 42 days after the last dose of the prior study treatment until a second PD event, clinical deterioration, and/or intolerance to the crossover treatment for up to a maximum of 1 year (maximum 17 cycles on an every-21-day schedule).
- Total: Total of all reporting groups
Arm/Group | Arm A (FL+DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm B (FL+DLBCL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Cohort C (FL): RTX + Polatuzumab | Cohort E (FL+DLBCL): Obinutuzumab + Polatuzumab | Cohort G (Expansion, FL): Obinutuzumab + Polatuzumab | Cohort H (Expansion, DLBCL): Obinutuzumab + Polatuzumab | Total
Number analyzed (Participants) | 63 | 59 | 20 | 9 | 40 | 40 | 231
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 29 | 25 | 12 | 4 | 23 | 16 | 109
  >=65 years | 34 | 34 | 8 | 5 | 17 | 24 | 122
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 24 | 8 | 2 | 16 | 18 | 95
  Male | 36 | 35 | 12 | 7 | 24 | 22 | 136
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 5 | 1 | 0 | 0 | 2 | 10
  Not Hispanic or Latino | 48 | 44 | 19 | 9 | 33 | 36 | 189
  Unknown or Not Reported | 13 | 10 | 0 | 0 | 7 | 2 | 32

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Best Overall Response (OR) of Complete Response (CR) or Partial Response (PR) as Determined by Modified Response and Progression Criteria for NHL: Rituximab Containing Regimens (Arms A and B, Cohort C)
Description: Tumor response was evaluated according to modified response and progression criteria for NHL published by Cheson et al (2007 and 2014) and confirmed by repeat assessments greater than or equal to (>/=) 4 weeks after initial documentation. CR was defined as disappearance of all clinical/radiographic evidence of disease, regression of lymph nodes to normal size, absence of splenomegaly, and absence of bone marrow involvement. PR was defined as >/=50 percent (%) decrease in sum of the products of greatest diameters (SPD) of up to six of the largest dominant lymph nodes, no increase in size of other nodes, liver, or spleen volume, a >/=50% decrease in SPD of hepatic and splenic nodules, absence of other organ involvement, and no new sites of disease. Participants with insufficient data to determine response were classified as non-responders.
Time Frame: Baseline up to 12 months after the last dose of study treatment (up to approximately 3.5 years)
Population: Rituximab Containing Regimens (Arms A and B, Cohort C): Analysis was performed on efficacy-evaluable population, which included all participants with baseline measurable disease and at least one post-baseline tumor assessment after study treatment.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Arm A (DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab: Participants with r/r DLBCL received RTX at a dose of 375 mg/m^2 administered via IV infusion on Day 1 and pinatuzumab vedotin at a dose of 2.4 mg/kg administered via IV infusion on Day 2 for the first 2 cycles. RTX and pinatuzumab were administered on the same day (Day 1) in subsequent cycles beginning with the third cycle, in the absence of any infusion-related adverse events. Participants who developed PD were treated with RTX at 375 mg/m^2 and polatuzumab vedotin at 2.4 mg/kg via IV infusion on Day 1, beginning no later than 42 days after the last dose of the prior study treatment until a second PD event, clinical deterioration, and/or intolerance to the crossover treatment for up to a maximum of 1 year (maximum 17 cycles on an every-21-day schedule).
- Arm A (FL): RTX+Pinatuzumab,Then RTX+Polatuzumab: Participants with r/r FL received RTX at a dose of 375 mg/m^2 administered via IV infusion on Day 1 and pinatuzumab vedotin at a dose of 2.4 mg/kg administered via IV infusion on Day 2 for the first 2 cycles. RTX and pinatuzumab were administered on the same day (Day 1) in subsequent cycles beginning with the third cycle, in the absence of any infusion-related adverse events. Participants who developed PD were treated with RTX at 375 mg/m^2 and polatuzumab vedotin at 2.4 mg/kg via IV infusion on Day 1, beginning no later than 42 days after the last dose of the prior study treatment until a second PD event, clinical deterioration, and/or intolerance to the crossover treatment for up to a maximum of 1 year (maximum 17 cycles on an every-21-day schedule).
- Arm B (DLBCL): RTX+Polatuzumab,Then RTX+Pinatuzumab: Participants with r/r DLBCL received RTX at a dose of 375 mg/m^2 administered via IV infusion on Day 1 and polatuzumab vedotin at a dose of 2.4 mg/kg administered via IV infusion on Day 2 for the first 2 cycles. RTX and polatuzumab were administered on the same day (Day 1) in subsequent cycles beginning with the third cycle, in the absence of any infusion-related adverse events. Participants who developed PD were treated with RTX at 375 mg/m^2 and pinatuzumab vedotin at 2.4 mg/kg via IV infusion on Day 1, beginning no later than 42 days after the last dose of the prior study treatment until a second PD event, clinical deterioration, and/or intolerance to the crossover treatment for up to a maximum of 1 year (maximum 17 cycles on an every-21-day schedule).
- Arm B (FL): RTX+Polatuzumab,Then RTX+Pinatuzumab: Participants with r/r FL received RTX at a dose of 375 mg/m^2 administered via IV infusion on Day 1 and polatuzumab vedotin at a dose of 2.4 mg/kg administered via IV infusion on Day 2 for the first 2 cycles. RTX and polatuzumab were administered on the same day (Day 1) in subsequent cycles beginning with the third cycle, in the absence of any infusion-related adverse events. Participants who developed PD were treated with RTX at 375 mg/m^2 and pinatuzumab vedotin at 2.4 mg/kg via IV infusion on Day 1, beginning no later than 42 days after the last dose of the prior study treatment until a second PD event, clinical deterioration, and/or intolerance to the crossover treatment for up to a maximum of 1 year (maximum 17 cycles on an every-21-day schedule).
Arm/Group | Arm A (DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm A (FL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm B (DLBCL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Arm B (FL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Cohort C (FL): RTX + Polatuzumab
Number analyzed (Participants) | 42 | 21 | 39 | 20 | 20
percentage of participants | 59.5 [45.67 to 72.32] | 61.9 [41.72 to 79.43] | 53.8 [39.58 to 67.65] | 70.0 [49.22 to 86.04] | 75.0 [54.44 to 89.59]

2. Primary Outcome: Duration of Objective Response (DOR) as Determined by Modified Response and Progression Criteria for NHL: Rituximab Containing Regimens (Arms A and B, Cohort C)
Description: Tumor response was evaluated according to modified response and progression criteria for NHL published by Cheson et al (2007 and 2014). DOR was defined as the time from the initial documentation of a CR or PR to the time of PD or death. CR was defined as disappearance of all clinical/radiographic evidence of disease, regression of lymph nodes to normal size, absence of splenomegaly, and absence of bone marrow involvement. PR was defined as >/=50% decrease in SPD of up to six of the largest dominant lymph nodes, no increase in size of other nodes, liver, or spleen volume, a >/=50% decrease in SPD of hepatic and splenic nodules, absence of other organ involvement, and no new sites of disease. PD was defined as appearance of any new lesion more than 1.5 centimeters (cm) in any axis, at least a 50% increase from nadir in the SPD or longest diameter of any previous lesion or node.
Time Frame: First occurrence of objective response up to PD/relapse or death due to any cause, whichever occurred first (up to approximately 3.5 years)
Population: Rituximab Containing Regimens (Arms A and B, Cohort C): Analysis was performed on efficacy-evaluable population participants who achieved objective response.
Measure: Median (Full Range); unit: months
Arm/Group | Arm A (DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm A (FL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm B (DLBCL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Arm B (FL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Cohort C (FL): RTX + Polatuzumab
Number analyzed (Participants) | 25 | 13 | 21 | 14 | 15
months | 6.24 [0.89 to 22.57] | 6.47 [0.03 to 23.52] | 13.37 [0.03 to 35.68] | 9.36 [0.03 to 19.35] | 12.85 [0.03 to 22.11]

3. Primary Outcome: Percentage of Participants With CR at End of Treatment (EOT) Based on Positron Emission Tomographic/Computed Tomography (PET/CT) Assessment Determined by Independent Review Committee (IRC) Per Lugano 2014 Response Criteria: Cohorts E, G, and H
Description: Tumor response assessment was performed by an IRC according to modified Lugano classification using PET/CT scan. CR was defined as a score of 1 (no uptake above background), 2 (uptake less than or equal to [</=] mediastinum), or 3 (uptake less than [<] mediastinum but </=liver) with or without a residual mass on PET 5-point scale (5-PS), for lymph nodes and extralymphatic sites; no new lesions; no evidence of fluorodeoxyglucose (FDG)-avid disease in bone marrow; and normal/immunohistochemistry (IHC)-negative bone marrow morphology. 90% confidence interval (CI) for percentage of responders was calculated using Clopper-Pearson method.
Time Frame: 6-8 weeks after Cycle 8 Day 1 (cycle length = 21 Days) or last study treatment (maximum up to 27-29 weeks)
Population: Obinutuzumab-Containing Cohorts (Cohorts E, G, and H): Analysis was performed on efficacy-evaluable population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants evaluable for this outcome measure.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Cohort E (DLBCL): Obinutuzumab + Polatuzumab: Participants with r/r DLBCL received obinutuzumab via IV infusion on Days 1, 8, 15 and polatuzumab vedotin at a dose of 1.8 mg/kg administered via IV infusion on Day 2 for the first cycle. In the absence of any infusion-related adverse events, obinutuzumab and polatuzumab vedotin were administered on the same day (Day 1) in subsequent cycles beginning with the second cycle for up to a maximum of 8 cycles or significant toxicity, disease progression, or withdrawal from study.
- Cohort E (FL): Obinutuzumab + Polatuzumab: Participants with r/r FL received obinutuzumab via IV infusion on Days 1, 8, 15 and polatuzumab vedotin at a dose of 1.8 mg/kg administered via IV infusion on Day 2 for the first cycle. In the absence of any infusion-related adverse events, obinutuzumab and polatuzumab vedotin were administered on the same day (Day 1) in subsequent cycles beginning with the second cycle for up to a maximum of 8 cycles or significant toxicity, disease progression, or withdrawal from study.
Arm/Group | Cohort E (DLBCL): Obinutuzumab + Polatuzumab | Cohort E (FL): Obinutuzumab + Polatuzumab | Cohort G (Expansion, FL): Obinutuzumab + Polatuzumab | Cohort H (Expansion, DLBCL): Obinutuzumab + Polatuzumab
Number analyzed (Participants) | 4 | 2 | 34 | 27
percentage of participants | 0 [0.00 to 52.71] | 50.0 [2.53 to 97.47] | 35.3 [21.79 to 50.82] | 0 [0.00 to 10.50]

4. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADA) to Pinatuzumab Vedotin
Description: Participants provided blood samples for evaluation of ADA. The number of participants with positive results for ADA against pinatuzumab vedotin at Baseline and at any of the post-baseline assessment time-points (overall 1.5 years) was reported. Participants positive at any post-baseline time points were post-baseline evaluable participants determined to have "Treatment-induced ADAs" or "Treatment-enhanced ADA" during the study period. Treatment-induced ADA = a participant with negative or missing Baseline ADA result(s) and at least one positive post-Baseline ADA result. Treatment-enhanced ADA = a participant with positive ADA result at Baseline who has one or more post Baseline titer results that are at least 0.60 titer unit greater than the Baseline titer result.
Time Frame: Baseline, post-baseline (up to approximately 5.5 years)
Population: Analysis was performed on safety-evaluable population (only participants who received pinatuzumab vedotin). Here, 'Overall Number of Participants Analyzed' signifies the number of participants evaluable for this outcome measure and 'Number Analyzed' signifies the number of participants evaluable at specified time points.
Measure: Number; unit: participants
Groups:
- Arm A (FL+DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab: Participants with r/r FL and DLBCL received RTX at a dose of 375 mg/m^2 administered via IV infusion on Day 1 and pinatuzumab vedotin at a dose of 2.4 mg/kg administered via IV infusion on Day 2 for the first 2 cycles. RTX and pinatuzumab were administered on the same day (Day 1) in subsequent cycles beginning with the third cycle, in the absence of any infusion-related adverse events. Participants who developed PD were treated with RTX at 375 mg/m^2 and polatuzumab vedotin at 2.4 mg/kg via IV infusion on Day 1, beginning no later than 42 days after the last dose of the prior study treatment until a second PD event, clinical deterioration, and/or intolerance to the crossover treatment for up to a maximum of 1 year (maximum 17 cycles on an every-21-day schedule).
Arm/Group | Arm A (FL+DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm B (FL+DLBCL): RTX+Polatuzumab,Then RTX+Pinatuzumab
Number analyzed (Participants) | 60 | 1
participants
  Baseline: number analyzed (Participants) | 60 | 0
  Baseline | 2 |
  Post-baseline: number analyzed (Participants) | 56 | 1
  Post-baseline | 0 | 0

5. Secondary Outcome: Number of Participants With ADA to Polatuzumab Vedotin
Description: Participants provided blood samples for evaluation of ADA. The number of participants with positive results for ADA against polatuzumab vedotin at Baseline and at any of the post-baseline assessment time-points (overall 1.5 years) was reported. Participants positive at any post-baseline time points were post-baseline evaluable participants determined to have "Treatment-induced ADAs" or "Treatment-enhanced ADA" during the study period. Treatment-induced ADA = a participant with negative or missing Baseline ADA result(s) and at least one positive post-Baseline ADA result. Treatment-enhanced ADA = a participant with positive ADA result at Baseline who has one or more post Baseline titer results that are at least 0.60 titer unit greater than the Baseline titer result.
Time Frame: Baseline, post-baseline (up to approximately 5.5 years)
Population: Analysis was performed on safety-evaluable population (only participants who received polatuzumab vedotin). Here, 'Overall Number of Participants Analyzed' signifies the number of participants evaluable for this outcome measure and 'Number Analyzed' signifies the number of participants evaluable at specified time points.
Measure: Number; unit: participants
Arm/Group | Arm A (FL+DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm B (FL+DLBCL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Cohort C (FL): RTX + Polatuzumab | Cohort E (FL+DLBCL): Obinutuzumab + Polatuzumab | Cohort G (Expansion, FL): Obinutuzumab + Polatuzumab | Cohort H (Expansion, DLBCL): Obinutuzumab + Polatuzumab
Number analyzed (Participants) | 2 | 59 | 20 | 8 | 37 | 36
participants
  Baseline: number analyzed (Participants) | 0 | 59 | 20 | 8 | 37 | 36
  Baseline |  | 1 | 0 | 0 | 0 | 0
  Post-baseline: number analyzed (Participants) | 2 | 53 | 20 | 6 | 36 | 36
  Post-baseline | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With ADA to Obinutuzumab
Description: Participants provided blood samples for evaluation of ADA. The number of participants with positive results for ADA against obinutuzumab at Baseline and at any of the post-baseline assessment time-points (overall 1.5 years) was reported. Participants positive at any post-baseline time points were post-baseline evaluable participants determined to have "Treatment-induced ADAs" or "Treatment-enhanced ADA" during the study period. Treatment-induced ADA = a participant with negative or missing Baseline ADA result(s) and at least one positive post-Baseline ADA result. Treatment-enhanced ADA = a participant with positive ADA result at Baseline who has one or more post Baseline titer results that are at least 0.60 titer unit greater than the Baseline titer result.
Time Frame: Baseline, post-baseline (up to approximately 5.5 years)
Population: Analysis was performed on safety-evaluable population (only participants who received obinutuzumab). Here, 'Overall Number of Participants Analyzed' signifies the number of participants evaluable for this outcome measure and 'Number Analyzed' signifies the number of participants evaluable at specified time points.
Measure: Number; unit: participants
Arm/Group | Cohort E (FL+DLBCL): Obinutuzumab + Polatuzumab | Cohort G (Expansion, FL): Obinutuzumab + Polatuzumab | Cohort H (Expansion, DLBCL): Obinutuzumab + Polatuzumab
Number analyzed (Participants) | 9 | 37 | 39
participants
  Baseline | 1 | 2 | 0
  Post-baseline: number analyzed (Participants) | 6 | 36 | 37
  Post-baseline | 0 | 0 | 0

7. Secondary Outcome: Percentage of Participants With PD as Determined by Modified Response and Progression Criteria for NHL or Death Due to Any Cause: Rituximab Containing Regimens (Arms A and B, Cohort C)
Description: Tumor response was evaluated according to modified response and progression criteria for NHL published by Cheson et al (2007 and 2014) and confirmed by repeat assessments >/=4 weeks after initial documentation. PD was defined as appearance of any new lesion more than 1.5 cm in any axis, at least a 50% increase from nadir in the SPD or longest diameter of any previous lesion or node.
Time Frame: Baseline up to PD or death due to any cause, whichever occurred first (up to approximately 5.5 years)
Population: Rituximab Containing Regimens (Arms A and B, Cohort C): Analysis was performed on efficacy-evaluable population.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A (DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm A (FL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm B (DLBCL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Arm B (FL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Cohort C (FL): RTX + Polatuzumab
Number analyzed (Participants) | 42 | 21 | 39 | 20 | 20
percentage of participants | 85.7 | 52.4 | 76.9 | 55.0 | 60.0

8. Secondary Outcome: Progression-free Survival (PFS) as Determined by Modified Response and Progression Criteria for NHL: Rituximab Containing Regimens (Arms A and B, Cohort C)
Description: Tumor response was evaluated according to modified response and progression criteria for NHL published by Cheson et al (2007 and 2014) and confirmed by repeat assessments >/=4 weeks after initial documentation. PD was defined as appearance of any new lesion more than 1.5 cm in any axis, at least a 50% increase from nadir in the SPD or longest diameter of any previous lesion or node. PFS was defined as the time from the date of randomization to the date of PD or death from any cause, whichever occurred first. In absence of PD or death, PFS was censored at the date of the last tumor assessment. Participants with no post-baseline tumor assessment were censored on the date of randomization or date of enrollment. The median PFS was estimated using Kaplan-Meier estimates and the 95% CI for median was computed using the method of Brookmeyer and Crowley.
Time Frame: Baseline up to PD or death due to any cause, whichever occurred first (up to approximately 5.5 years)
Population: Rituximab Containing Regimens (Arms A and B, Cohort C): Analysis was performed on efficacy-evaluable population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm A (FL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm B (DLBCL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Arm B (FL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Cohort C (FL): RTX + Polatuzumab
Number analyzed (Participants) | 42 | 21 | 39 | 20 | 20
months | 5.388 [3.943 to 10.579] | 12.682 [8.936 to 27.466] | 5.552 [4.304 to 12.780] | 15.277 [12.189 to 25.133] | 18.103 [11.598 to 30.259]

9. Secondary Outcome: Percentage of Participants Who Died Due to Any Cause: Rituximab Containing Regimens (Arms A and B, Cohort C)
Description: Percentage of participants who died due to any cause was reported.
Time Frame: Baseline up to death due to any cause (from baseline up to study completion date, up to approximately 5.5 years)
Population: Rituximab Containing Regimens (Arms A and B, Cohort C): Analysis was performed on efficacy-evaluable population.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A (DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm A (FL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm B (DLBCL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Arm B (FL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Cohort C (FL): RTX + Polatuzumab
Number analyzed (Participants) | 42 | 21 | 39 | 20 | 20
percentage of participants | 66.7 | 23.8 | 61.5 | 15.0 | 20.0

10. Secondary Outcome: Overall Survival (OS): Rituximab Containing Regimens (Arms A and B, Cohort C)
Description: OS was defined as the time from the date of randomization or enrollment to the date of death from any cause. The median OS was estimated using Kaplan-Meier estimates and the 95% CI for median was computed using the method of Brookmeyer and Crowley.
Time Frame: Baseline up to death due to any cause (from baseline up to study completion date, up to approximately 5.5 years)
Population: Rituximab Containing Regimens (Arms A and B, Cohort C): Analysis was performed on efficacy-evaluable population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A (DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm A (FL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm B (DLBCL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Arm B (FL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Cohort C (FL): RTX + Polatuzumab
Number analyzed (Participants) | 42 | 21 | 39 | 20 | 20
months | 16.493 [7.458 to 32.460] | NA [44.025 to NA] — Median and Upper Limit of CI could not be estimated because very few participants (<50%) had the event of interest. | 18.760 [10.415 to 38.571] | NA [NA to NA] — Median and corresponding CI could not be estimated because very few participants (<50%) had the event of interest. | NA [NA to NA] — Median and corresponding CI could not be estimated because very few participants (<50%) had the event of interest.

11. Secondary Outcome: Percentage of Participants With CR at EOT Based on PET/CT Assessment as Determined by Investigator Per Lugano 2014 Response Criteria: Obinutuzumab-Containing Cohorts (Cohorts E, G, and H)
Description: Tumor response assessment was performed by the investigator according to modified Lugano classification using PET/CT scan. CR was defined as a score of 1 (no uptake above background), 2 (uptake </=mediastinum), or 3 (uptake <mediastinum but </=liver) with or without a residual mass on PET 5-PS, for lymph nodes and extralymphatic sites; no new lesions; no evidence of FDG-avid disease in bone marrow; and normal/IHC-negative bone marrow morphology. 90% CI for percentage of responders was calculated using Clopper-Pearson method.
Time Frame: 6-8 weeks after Cycle 8 Day 1 (cycle length = 21 Days) or last study treatment (maximum up to 27-29 weeks)
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort E (DLBCL): Obinutuzumab + Polatuzumab | Cohort E (FL): Obinutuzumab + Polatuzumab | Cohort G (Expansion, FL): Obinutuzumab + Polatuzumab | Cohort H (Expansion, DLBCL): Obinutuzumab + Polatuzumab
Number analyzed (Participants) | 4 | 3 | 36 | 33
percentage of participants | 25.0 [1.27 to 75.14] | 66.7 [13.54 to 98.30] | 33.3 [20.49 to 48.34] | 15.2 [6.17 to 29.25]

12. Secondary Outcome: Percentage of Participants With OR at EOT Based on PET/CT Assessment as Determined by IRC Per Lugano 2014 Response Criteria: Obinutuzumab-Containing Cohorts (Cohorts E, G, and H)
Description: Tumor response assessment was performed by an IRC according to modified Lugano classification using PET/CT scan. OR was defined as a response of CR or PR. CR was defined as a score of 1 (no uptake above background), 2 (uptake </=mediastinum), or 3 (uptake <mediastinum but </=liver) with or without a residual mass on PET 5-PS, for lymph nodes and extralymphatic sites; no new lesions; no evidence of FDG-avid disease in bone marrow; and normal/IHC-negative bone marrow morphology. PR was defined as a score 4 (uptake moderately greater than [>] liver) or 5 (uptake markedly >liver and/or new lesions) with reduced uptake compared with baseline and residual mass(es) of any size on PET 5-PS for lymph nodes and extralymphatic sites; no new lesions; and reduced residual uptake in bone marrow compared with baseline. 90% CI for percentage of responders was calculated using Clopper-Pearson method.
Time Frame: 6-8 weeks after Cycle 8 Day 1 (cycle length = 21 Days) or last study treatment (maximum up to 27-29 weeks)
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort E (DLBCL): Obinutuzumab + Polatuzumab | Cohort E (FL): Obinutuzumab + Polatuzumab | Cohort G (Expansion, FL): Obinutuzumab + Polatuzumab | Cohort H (Expansion, DLBCL): Obinutuzumab + Polatuzumab
Number analyzed (Participants) | 4 | 2 | 34 | 27
percentage of participants | 25.0 [1.27 to 75.14] | 100.0 [22.36 to 100.00] | 64.7 [49.18 to 78.21] | 18.5 [7.59 to 35.06]

13. Secondary Outcome: Percentage of Participants With OR at EOT Based on PET/CT Assessment as Determined by the Investigator Per Lugano 2014 Response Criteria: Obinutuzumab-Containing Cohorts (Cohorts E, G, and H)
Description: Tumor response assessment was performed by investigator according to modified Lugano classification using PET/CT scan. OR was defined as a response of CR or PR. CR was defined as a score of 1 (no uptake above background), 2 (uptake </=mediastinum), or 3 (uptake <mediastinum but </=liver) with or without a residual mass on PET 5-PS, for lymph nodes and extralymphatic sites; no new lesions; no evidence of FDG-avid disease in bone marrow; and normal/IHC-negative bone marrow morphology. PR was defined as a score 4 (uptake moderately >liver) or 5 (uptake markedly >liver and/or new lesions) with reduced uptake compared with baseline and residual mass(es) of any size on PET 5-PS for lymph nodes and extralymphatic sites; no new lesions; and reduced residual uptake in bone marrow compared with baseline. 90% CI for percentage of responders was calculated using Clopper-Pearson method.
Time Frame: 6-8 weeks after Cycle 8 Day 1 (cycle length = 21 Days) or last study treatment (maximum up to 27-29 weeks)
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort E (DLBCL): Obinutuzumab + Polatuzumab | Cohort E (FL): Obinutuzumab + Polatuzumab | Cohort G (Expansion, FL): Obinutuzumab + Polatuzumab | Cohort H (Expansion, DLBCL): Obinutuzumab + Polatuzumab
Number analyzed (Participants) | 4 | 3 | 36 | 33
percentage of participants | 25.0 [1.27 to 75.14] | 66.7 [13.54 to 98.30] | 63.9 [48.83 to 77.15] | 21.2 [10.40 to 36.18]

14. Secondary Outcome: Percentage of Participants With CR at EOT Based on CT Assessment Alone as Determined by IRC Per Lugano 2014 Response Criteria: Obinutuzumab-Containing Cohorts (Cohorts E + H and E + G)
Description: Tumor response assessment was performed by an IRC according to modified Lugano classification using CT scan. CR was defined as reduction of longest transverse diameter (LDi) of target nodes/nodal masses to less than or equal to (</=) 1.5 cm, no extralymphatic sites of disease, absence of non-measured lesions and new lesions, reduction of enlarged organs to normal, and normal/IHC-negative bone marrow morphology. 90% CI for percentage of responders was calculated using Clopper-Pearson method.
Time Frame: 6-8 weeks after Cycle 8 Day 1 (cycle length = 21 Days) or last study treatment (maximum up to 27-29 weeks)
Population: Obinutuzumab-Containing Cohorts (Cohorts E + H and E + G): Analysis was performed on efficacy-evaluable population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants evaluable for this outcome measure.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Cohort E + Cohort H (DLBCL): Obinutuzumab + Polatuzumab: Participants with r/r DLBCL received obinutuzumab at a dose of 1000 mg via IV infusion on Days 1, 8, 15 and polatuzumab vedotin at a dose of 1.8 mg/kg administered via IV infusion on Day 2 for the first cycle. In the absence of any infusion-related adverse events, obinutuzumab and polatuzumab vedotin were administered on the same day (Day 1) in subsequent cycles beginning with the second cycle for up to a maximum of 8 cycles or significant toxicity, disease progression, or withdrawal from study.
- Cohort E + Cohort G (FL): Obinutuzumab + Polatuzumab: Participants with r/r FL received obinutuzumab via IV infusion on Days 1, 8, 15 and polatuzumab vedotin at a dose of 1.8 mg/kg administered via IV infusion on Day 2 for the first cycle. In the absence of any infusion-related adverse events, obinutuzumab and polatuzumab vedotin were administered on the same day (Day 1) in subsequent cycles beginning with the second cycle for up to a maximum of 8 cycles or significant toxicity, disease progression, or withdrawal from study.
Arm/Group | Cohort E + Cohort H (DLBCL): Obinutuzumab + Polatuzumab | Cohort E + Cohort G (FL): Obinutuzumab + Polatuzumab
Number analyzed (Participants) | 31 | 36
percentage of participants | 6.5 [1.2 to 19.0] | 13.9 [5.6 to 27.0]

15. Secondary Outcome: Percentage of Participants With CR at EOT Based on CT Assessment Alone as Determined by Investigator Per Lugano 2014 Response Criteria: Obinutuzumab-Containing Cohorts (Cohorts E + H and E + G)
Description: Tumor response assessment was performed by investigator according to modified Lugano classification using CT scan. CR was defined as reduction of LDi of target nodes/nodal masses to </=1.5 cm, no extralymphatic sites of disease, absence of non-measured lesions and new lesions, reduction of enlarged organs to normal, and normal/IHC-negative bone marrow morphology. 90% CI for percentage of responders was calculated using Clopper-Pearson method.
Time Frame: 6-8 weeks after Cycle 8 Day 1 (cycle length = 21 Days) or last study treatment (maximum up to 27-29 weeks)
Population: as for outcome 14
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort E + Cohort H (DLBCL): Obinutuzumab + Polatuzumab | Cohort E + Cohort G (FL): Obinutuzumab + Polatuzumab
Number analyzed (Participants) | 37 | 39
percentage of participants | 10.8 [3.8 to 23.1] | 20.5 [10.6 to 34.0]

16. Secondary Outcome: Percentage of Participants With OR at EOT Based on CT Assessment Alone as Determined by IRC Per Lugano 2014 Response Criteria: Obinutuzumab-Containing Cohorts (Cohorts E + H and E + G)
Description: Tumor response assessment was performed by an IRC according to modified Lugano classification using CT scan. OR was defined as a response of CR or PR. CR was defined as reduction of LDi of target nodes/nodal masses to </=1.5 cm, no extralymphatic sites of disease, absence of non-measured lesions and new lesions, reduction of enlarged organs to normal, and normal/IHC-negative bone marrow morphology. PR was defined as >/=50% decrease in SPD of up to 6 target measurable nodes and extra-nodal sites; absence/reduction/no increase in size of non-measured lesions; reduction in length of spleen by at least >50% beyond normal; and no new lesions. 90% CI for percentage of responders was calculated using Clopper-Pearson method.
Time Frame: 6-8 weeks after Cycle 8 Day 1 (cycle length = 21 Days) or last study treatment (maximum up to 27-29 weeks)
Population: as for outcome 14
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort E + Cohort H (DLBCL): Obinutuzumab + Polatuzumab | Cohort E + Cohort G (FL): Obinutuzumab + Polatuzumab
Number analyzed (Participants) | 31 | 36
percentage of participants | 25.8 [13.5 to 41.8] | 66.7 [51.7 to 79.5]

17. Secondary Outcome: Percentage of Participants With OR at EOT Based on CT Assessment Alone as Determined by Investigator Per Lugano 2014 Response Criteria: Obinutuzumab-Containing Cohorts (Cohorts E + H and E + G)
Description: Tumor response assessment was performed by investigator according to modified Lugano classification using CT scan. OR was defined as a response of CR or PR. CR was defined as reduction of LDi of target nodes/nodal masses to </=1.5 cm, no extralymphatic sites of disease, absence of non-measured lesions and new lesions, reduction of enlarged organs to normal, and normal/IHC-negative bone marrow morphology. PR was defined as >/=50% decrease in SPD of up to 6 target measurable nodes and extra-nodal sites; absence/reduction/no increase in size of non-measured lesions; reduction in length of spleen by at least >50% beyond normal; and no new lesions. 90% CI for percentage of responders was calculated using Clopper-Pearson method.
Time Frame: 6-8 weeks after Cycle 8 Day 1 (cycle length = 21 Days) or last study treatment (maximum up to 27-29 weeks)
Population: as for outcome 14
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort E + Cohort H (DLBCL): Obinutuzumab + Polatuzumab | Cohort E + Cohort G (FL): Obinutuzumab + Polatuzumab
Number analyzed (Participants) | 37 | 39
percentage of participants | 21.6 [11.2 to 35.6] | 64.1 [49.7 to 76.8]

18. Secondary Outcome: Percentage of Participants With Best OR Based on PET/CT or CT Assessment as Determined by Investigator Per Lugano 2014 Response Criteria: Obinutuzumab-Containing Cohorts (Cohorts E, G, and H)
Description: Tumor response assessment was performed by investigator according to modified Lugano classification using PET/CT or CT scan. Best OR was defined as a response of CR or PR. CR was defined as a score of 1 (no uptake above background), 2 (uptake </=mediastinum), or 3 (uptake <mediastinum but </=liver) with or without a residual mass on PET 5-PS, for lymph nodes and extralymphatic sites; no new lesions; no evidence of FDG-avid disease in bone marrow; and normal/IHC-negative bone marrow morphology. PR was defined as a score 4 (uptake moderately >liver) or 5 (uptake markedly >liver and/or new lesions) with reduced uptake compared with baseline and residual mass(es) of any size on PET 5-PS for lymph nodes and extralymphatic sites; no new lesions; and reduced residual uptake in bone marrow compared with baseline. 90% CI for percentage of responders was calculated using Clopper-Pearson method.
Time Frame: Baseline up to disease progression or death, whichever occurred first (up to approximately 5.5 years)
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort E (DLBCL): Obinutuzumab + Polatuzumab | Cohort E (FL): Obinutuzumab + Polatuzumab | Cohort G (Expansion, FL): Obinutuzumab + Polatuzumab | Cohort H (Expansion, DLBCL): Obinutuzumab + Polatuzumab
Number analyzed (Participants) | 5 | 4 | 39 | 39
percentage of participants | 20.0 [1.02 to 65.74] | 50.0 [9.76 to 90.24] | 74.4 [60.40 to 85.38] | 43.6 [30.00 to 57.94]

19. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to Infinity (AUCinf) of Rituximab: Rituximab Containing Regimens (Arms A and B, Cohort C)
Description: AUCinf for rituximab was estimated from serum concentration data using non-compartmental analysis.
Time Frame: Pre-infusion (Hour 0) & 30 minutes post-infusion (infusion length= 2-6 hours) on Day 1 of Cycle 1; Day 8, Day 15 of Cycle 1 (Cycle length= 21 days)
Population: Rituximab Containing Regimens (Arms A and B, Cohort C): Analysis was performed on all participants with measurable pharmacokinetic (PK) concentrations. Here, 'Overall Number of Participants Analyzed' signifies the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: day*micrograms (mcg)/milliliter (mL)
Arm/Group | Arm A (DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm A (FL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm B (DLBCL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Arm B (FL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Cohort C (FL): RTX + Polatuzumab
Number analyzed (Participants) | 25 | 15 | 26 | 11 | 15
day*micrograms (mcg)/milliliter (mL) | 5640 (8320) | 3350 (1180) | 4200 (2620) | 3910 (2480) | 2660 (879)

20. Secondary Outcome: Maximum Observed Concentration (Cmax) of Rituximab: Rituximab Containing Regimens (Arms A and B, Cohort C)
Description: Cmax for rituximab was estimated from serum concentration data using non-compartmental analysis.
Time Frame: as for outcome 19
Population: Rituximab Containing Regimens (Arms A and B, Cohort C): Analysis was performed on all participants with measurable PK concentrations. Here, 'Overall Number of Participants Analyzed' signifies the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Arm A (DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm A (FL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm B (DLBCL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Arm B (FL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Cohort C (FL): RTX + Polatuzumab
Number analyzed (Participants) | 36 | 18 | 35 | 16 | 18
mcg/mL | 217 (61.5) | 225 (40.9) | 232 (72.7) | 228 (83.3) | 227 (32.4)

21. Secondary Outcome: Systemic Clearance (CL) of Rituximab: Rituximab Containing Regimens (Arms A and B, Cohort C)
Description: CL for rituximab was estimated from serum concentration data using non-compartmental analysis.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mL/day/meter-square (m^2)
Arm/Group | Arm A (DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm A (FL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm B (DLBCL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Arm B (FL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Cohort C (FL): RTX + Polatuzumab
Number analyzed (Participants) | 25 | 15 | 26 | 11 | 15
mL/day/meter-square (m^2) | 113.97 (61.41) | 124.53 (41.12) | 116.26 (59.99) | 134.31 (97.45) | 158.57 (60.47)

22. Secondary Outcome: Half-Life (t1/2) of Rituximab: Rituximab Containing Regimens (Arms A and B, Cohort C)
Description: t1/2 for rituximab was estimated from serum concentration data using non-compartmental analysis.
  Time Frame: Pre-infusion (Hour 0) & 30 minutes post-infusion (infusion length= 2-6 hours) on Day 1 of Cycle 1-4 and every 4th Cycle thereafter (approximately up to 1.5 years); Day 8, Day 15 of Cycle 1 and 3; 30 Days after last infusion; 2, 4, & 6 months after treatment completion visit (approximately up to 1.5 years, Cycle length= 21 days).
Time Frame: Day 1 up to 1.5 years (detailed timeframe is provided in the Outcome Measure Description)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm A (DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm A (FL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm B (DLBCL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Arm B (FL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Cohort C (FL): RTX + Polatuzumab
Number analyzed (Participants) | 25 | 15 | 26 | 11 | 15
days | 35.3 (56.3) | 18.7 (6.23) | 25.6 (18.0) | 19.8 (7.34) | 14.4 (3.62)

23. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Rituximab: Rituximab Containing Regimens (Arms A and B, Cohort C)
Description: Vss for rituximab was estimated from serum concentration data using non-compartmental analysis.
  Time Frame: Pre-infusion (Hour 0) & 30 minutes post-infusion (infusion length= 2-6 hours) on Day 1 of Cycle 1-4 and every 4th Cycle thereafter (approximately up to 1.5 years); Day 8, Day 15 of Cycle 1 and 3; 30 Days after last infusion; 2, 4, & 6 months after treatment completion visit (approximately up to 1.5 years, Cycle length= 21 days)
Time Frame: Day 1 up to 1.5 years (detailed timeframe is provided in the Outcome Measure Description)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: mL/m^2
Arm/Group | Arm A (DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm A (FL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm B (DLBCL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Arm B (FL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Cohort C (FL): RTX + Polatuzumab
Number analyzed (Participants) | 25 | 15 | 26 | 11 | 15
mL/m^2 | 2901.85 (1009.31) | 2802.96 (678.33) | 2988.90 (788.89) | 2839.26 (730.10) | 2654.46 (413.19)

24. Secondary Outcome: AUCinf of Total Antibody for Pinatuzumab Vedotin at Dose Level 2.4 mg/kg Given in Combination With Rituximab
Description: AUCinf of total antibody for pinatuzumab vedotin was estimated from serum concentration data using non-compartmental analysis. Total antibody is defined as antibody with Monomethyl Auristatin E (MMAE)-to-antibody ratio equal or greater than zero, including fully conjugated, partially unconjugated, and fully unconjugated antibody.
Time Frame: Pre-infusion (Hour 0) & 30 minutes Post-infusion (infusion length=30-90 minutes) on Day 1 of Cycle 1; Day 8, Day 15 of Cycle 1 (Cycle length= 21 Days)
Population: Analysis was performed on all participants who received pinatuzumab vedotin (Arm A) with measurable PK concentrations. Here, 'Overall Number of Participants Analyzed' signifies the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: day*mcg/mL
Arm/Group | Arm A (DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm A (FL): RTX+Pinatuzumab,Then RTX+Polatuzumab
Number analyzed (Participants) | 27 | 15
day*mcg/mL | 309 (67.7) | 315 (111)

25. Secondary Outcome: AUCinf of Antibody Conjugated Monomethyl Auristatin E (acMMAE) for Pinatuzumab Vedotin at Dose Level 2.4 mg/kg Given in Combination With Rituximab
Description: AUCinf of acMMAE for pinatuzumab was estimated from plasma concentration data using non-compartmental analysis. Antibody conjugated MMAE is the total concentration of MMAE that was conjugated to the antibody.
Time Frame: as for outcome 24
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: day*nanogram (ng)/mL
Arm/Group | Arm A (DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm A (FL): RTX+Pinatuzumab,Then RTX+Polatuzumab
Number analyzed (Participants) | 39 | 17
day*nanogram (ng)/mL | 2840 (555) | 3110 (828)

26. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero To Last Measurable Concentration (AUClast) of Unconjugated MMAE for Pinatuzumab Vedotin at Dose Level 2.4 mg/kg Given in Combination With Rituximab
Description: AUClast of unconjugated MMAE was estimated from plasma concentration data using non-compartmental analysis. Unconjugated MMAE is the total concentration of MMAE that was not conjugated to the antibody.
Time Frame: as for outcome 24
Population: Analysis was performed on all participants who received pinatuzumab vedotin (Arm A) with measurable PK concentrations.
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Arm A (DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm A (FL): RTX+Pinatuzumab,Then RTX+Polatuzumab
Number analyzed (Participants) | 39 | 21
day*ng/mL | 34.2 (24.0) | 33.5 (17.5)

27. Secondary Outcome: Cmax of Total Antibody for Pinatuzumab Vedotin at Dose Level 2.4 mg/kg Given in Combination With Rituximab
Description: Cmax of total antibody for pinatuzumab vedotin was estimated from serum concentration data using non-compartmental analysis. Total antibody is defined as antibody with MMAE-to-antibody ratio equal or greater than zero, including fully conjugated, partially unconjugated, and fully unconjugated antibody.
Time Frame: as for outcome 24
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Arm A (DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm A (FL): RTX+Pinatuzumab,Then RTX+Polatuzumab
Number analyzed (Participants) | 39 | 20
mcg/mL | 42.5 (11.6) | 48.3 (9.34)

28. Secondary Outcome: Cmax of acMMAE for Pinatuzumab Vedotin at Dose Level 2.4 mg/kg Given in Combination With Rituximab
Description: Cmax of acMMAE for pinatuzumab was estimated from plasma concentration data using non-compartmental analysis. acMMAE is the total concentration of MMAE that was conjugated to the antibody.
Time Frame: as for outcome 24
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm A (DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm A (FL): RTX+Pinatuzumab,Then RTX+Polatuzumab
Number analyzed (Participants) | 38 | 21
ng/mL | 850 (222) | 994 (190)

29. Secondary Outcome: Cmax of Unconjugated MMAE for Pinatuzumab Vedotin at Dose Level 2.4 mg/kg Given in Combination With Rituximab
Description: Cmax of unconjugated MMAE was estimated from plasma concentration data using non-compartmental analysis. Unconjugated MMAE is the total concentration of MMAE that was not conjugated to the antibody.
Time Frame: as for outcome 24
Population: Analysis was performed on all participants who received pinatuzumab vedotin (Arm A) with measurable PK concentrations.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm A (DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm A (FL): RTX+Pinatuzumab,Then RTX+Polatuzumab
Number analyzed (Participants) | 39 | 21
ng/mL | 4.39 (3.15) | 4.20 (2.32)

30. Secondary Outcome: AUCinf of Total Antibody for Polatuzumab Vedotin at Dose Level 2.4 mg/kg Given in Combination With Rituximab
Description: AUCinf of total antibody for polatuzumab vedotin was estimated from serum concentration data using non-compartmental analysis. Total antibody is defined as antibody with MMAE-to-antibody ratio equal or greater than zero, including fully conjugated, partially unconjugated, and fully unconjugated antibody.
Time Frame: as for outcome 24
Population: Analysis was performed on all participants who received polatuzumab vedotin at dose level 2.4 mg/kg in combination with rituximab (Arm B) with measurable PK concentrations. Here, 'Overall Number of Participants Analyzed' signifies the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: day*mcg/mL
Arm/Group | Arm B (DLBCL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Arm B (FL): RTX+Polatuzumab,Then RTX+Pinatuzumab
Number analyzed (Participants) | 26 | 17
day*mcg/mL | 412 (108) | 428 (106)

31. Secondary Outcome: AUCinf of acMMAE for Polatuzumab Vedotin at Dose Level 2.4 mg/kg Given in Combination With Rituximab
Description: AUCinf of acMMAE for polatuzumab vedotin was estimated from plasma concentration data using non-compartmental analysis. acMMAE is the total concentration of MMAE that was conjugated to the antibody.
Time Frame: as for outcome 24
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Arm B (DLBCL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Arm B (FL): RTX+Polatuzumab,Then RTX+Pinatuzumab
Number analyzed (Participants) | 30 | 17
day*ng/mL | 3660 (843) | 3510 (1160)

32. Secondary Outcome: AUClast of Unconjugated MMAE for Polatuzumab Vedotin at Dose Level 2.4 mg/kg Given in Combination With Rituximab
Description: AUClast of Unconjugated MMAE for polatuzumab vedotin was estimated from plasma concentration data using non-compartmental analysis. Unconjugated MMAE is the total concentration of MMAE that was not conjugated to the antibody.
Time Frame: as for outcome 24
Population: Analysis was performed on all participants who received polatuzumab vedotin at dose level 2.4 mg/kg in combination with rituximab (Arm B) with measurable PK concentrations.
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Arm B (DLBCL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Arm B (FL): RTX+Polatuzumab,Then RTX+Pinatuzumab
Number analyzed (Participants) | 39 | 18
day*ng/mL | 31.7 (17.2) | 29.5 (25.0)

33. Secondary Outcome: Cmax of Total Antibody for Polatuzumab Vedotin at Dose Level 2.4 mg/kg Given in Combination With Rituximab
Description: Cmax of total antibody for polatuzumab vedotin was estimated from serum concentration data using non-compartmental analysis. Total antibody is defined as antibody with MMAE-to-antibody ratio equal or greater than zero, including fully conjugated, partially unconjugated, and fully unconjugated antibody.
Time Frame: as for outcome 24
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Arm B (DLBCL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Arm B (FL): RTX+Polatuzumab,Then RTX+Pinatuzumab
Number analyzed (Participants) | 38 | 16
mcg/mL | 51.9 (12.3) | 55.9 (12.8)

34. Secondary Outcome: Cmax of acMMAE for Polatuzumab Vedotin at Dose Level 2.4 mg/kg Given in Combination With Rituximab
Description: Cmax of acMMAE for polatuzumab vedotin was estimated from plasma concentration data using non-compartmental analysis. acMMAE is the total concentration of MMAE that was conjugated to the antibody.
Time Frame: as for outcome 24
Population: as for outcome 30
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm B (DLBCL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Arm B (FL): RTX+Polatuzumab,Then RTX+Pinatuzumab
Number analyzed (Participants) | 38 | 17
ng/mL | 948 (204) | 968 (268)

35. Secondary Outcome: Cmax of Unconjugated MMAE for Polatuzumab Vedotin at Dose Level 2.4 mg/kg Given in Combination With Rituximab
Description: Cmax of Unconjugated MMAE for polatuzumab vedotin was estimated from plasma concentration data using non-compartmental analysis. Unconjugated MMAE is the total concentration of MMAE that was not conjugated to the antibody.
Time Frame: as for outcome 24
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Arm B (DLBCL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Arm B (FL): RTX+Polatuzumab,Then RTX+Pinatuzumab
Number analyzed (Participants) | 39 | 18
ng/mL | 3.72 (1.98) | 3.29 (2.71)

36. Secondary Outcome: AUCinf of Total Antibody for Polatuzumab Vedotin at Dose Level 1.8 mg/kg Given in Combination With Rituximab
Description: as for outcome 30
Time Frame: as for outcome 24
Population: Analysis was performed on all participants who received polatuzumab vedotin at dose level 1.8 mg/kg in combination with rituximab (Cohort C) with measurable PK concentrations. Here, 'Overall Number of Participants Analyzed' signifies the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: day*mcg/mL
Arm/Group | Cohort C (FL): RTX + Polatuzumab
Number analyzed (Participants) | 17
day*mcg/mL | 258 (84.1)

37. Secondary Outcome: AUCinf of acMMAE for Polatuzumab Vedotin at Dose Level 1.8 mg/kg Given in Combination With Rituximab
Description: as for outcome 31
Time Frame: as for outcome 24
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Cohort C (FL): RTX + Polatuzumab
Number analyzed (Participants) | 15
day*ng/mL | 2600 (630)

38. Secondary Outcome: AUClast of Unconjugated MMAE for Polatuzumab Vedotin at Dose Level 1.8 mg/kg Given in Combination With Rituximab
Description: as for outcome 32
Time Frame: as for outcome 24
Population: Analysis was performed on all participants who received polatuzumab vedotin at dose level 1.8 mg/kg in combination with rituximab (Cohort C) with measurable PK concentrations.
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Cohort C (FL): RTX + Polatuzumab
Number analyzed (Participants) | 20
day*ng/mL | 17.7 (9.39)

39. Secondary Outcome: Cmax of Total Antibody for Polatuzumab Vedotin at Dose Level 1.8 mg/kg Given in Combination With Rituximab
Description: as for outcome 33
Time Frame: as for outcome 24
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Cohort C (FL): RTX + Polatuzumab
Number analyzed (Participants) | 19
mcg/mL | 42.2 (7.92)

40. Secondary Outcome: Cmax of acMMAE for Polatuzumab Vedotin at Dose Level 1.8 mg/kg Given in Combination With Rituximab
Description: as for outcome 34
Time Frame: as for outcome 24
Population: as for outcome 36
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort C (FL): RTX + Polatuzumab
Number analyzed (Participants) | 17
ng/mL | 787 (113)

41. Secondary Outcome: Cmax of Unconjugated MMAE for Polatuzumab Vedotin at Dose Level 1.8 mg/kg Given in Combination With Rituximab
Description: as for outcome 35
Time Frame: as for outcome 24
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort C (FL): RTX + Polatuzumab
Number analyzed (Participants) | 20
ng/mL | 2.02 (1.34)

42. Secondary Outcome: AUCinf of Total Antibody for Polatuzumab Vedotin at Dose Level 1.8 mg/kg Given in Combination With Obinutuzumab
Description: as for outcome 30
Time Frame: as for outcome 24
Population: Analysis was performed on all participants who received polatuzumab vedotin at dose level 1.8 mg/kg in combination with obinutuzumab (Cohort E+H and E+G) with measurable PK concentrations. Here, 'Overall Number of Participants Analyzed' signifies the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: day*mcg/mL
Groups:
- Cohort E + Cohort G (FL): Obinutuzumab + Polatuzumab: Participants with r/r FL received obinutuzumab at a dose of 1000 mg via IV infusion on Days 1, 8, 15 and polatuzumab vedotin at a dose of 1.8 mg/kg administered via IV infusion on Day 2 for the first cycle. In the absence of any infusion-related adverse events, obinutuzumab and polatuzumab vedotin were administered on the same day (Day 1) in subsequent cycles beginning with the second cycle for up to a maximum of 8 cycles or significant toxicity, disease progression, or withdrawal from study.
Arm/Group | Cohort E + Cohort H (DLBCL): Obinutuzumab + Polatuzumab | Cohort E + Cohort G (FL): Obinutuzumab + Polatuzumab
Number analyzed (Participants) | 27 | 30
day*mcg/mL | 218 (89.1) | 215 (102)

43. Secondary Outcome: AUCinf of acMMAE for Polatuzumab Vedotin at Dose Level 1.8 mg/kg Given in Combination With Obinutuzumab
Description: as for outcome 31
Time Frame: as for outcome 24
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Cohort E + Cohort H (DLBCL): Obinutuzumab + Polatuzumab | Cohort E + Cohort G (FL): Obinutuzumab + Polatuzumab
Number analyzed (Participants) | 26 | 29
day*ng/mL | 2440 (665) | 2340 (875)

44. Secondary Outcome: AUClast of Unconjugated MMAE for Polatuzumab Vedotin at Dose Level 1.8 mg/kg Given in Combination With Obinutuzumab
Description: as for outcome 32
Time Frame: as for outcome 24
Population: Analysis was performed on all participants who received polatuzumab vedotin at dose level 1.8 mg/kg in combination with obinutuzumab (Cohort E+H and E+G) with measurable PK concentrations.
Measure: Mean (Standard Deviation); unit: day*ng/mL
Arm/Group | Cohort E + Cohort H (DLBCL): Obinutuzumab + Polatuzumab | Cohort E + Cohort G (FL): Obinutuzumab + Polatuzumab
Number analyzed (Participants) | 40 | 41
day*ng/mL | 27.9 (21.3) | 22.3 (9.46)

45. Secondary Outcome: Cmax of Total Antibody for Polatuzumab Vedotin at Dose Level 1.8 mg/kg Given in Combination With Obinutuzumab
Description: as for outcome 33
Time Frame: as for outcome 24
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Cohort E + Cohort H (DLBCL): Obinutuzumab + Polatuzumab | Cohort E + Cohort G (FL): Obinutuzumab + Polatuzumab
Number analyzed (Participants) | 37 | 38
mcg/mL | 35.0 (9.89) | 34.2 (7.89)

46. Secondary Outcome: Cmax of acMMAE for Polatuzumab Vedotin at Dose Level 1.8 mg/kg Given in Combination With Obinutuzumab
Description: as for outcome 34
Time Frame: as for outcome 24
Population: as for outcome 42
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort E + Cohort H (DLBCL): Obinutuzumab + Polatuzumab | Cohort E + Cohort G (FL): Obinutuzumab + Polatuzumab
Number analyzed (Participants) | 33 | 33
ng/mL | 711 (155) | 694 (161)

47. Secondary Outcome: Cmax of Unconjugated MMAE for Polatuzumab Vedotin at Dose Level 1.8 mg/kg Given in Combination With Obinutuzumab
Description: as for outcome 35
Time Frame: as for outcome 24
Population: as for outcome 44
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort E + Cohort H (DLBCL): Obinutuzumab + Polatuzumab | Cohort E + Cohort G (FL): Obinutuzumab + Polatuzumab
Number analyzed (Participants) | 40 | 41
ng/mL | 3.62 (3.73) | 2.80 (1.30)

48. Secondary Outcome: Cmax of Obinutuzumab: Obinutuzumab-Containing Cohorts (Cohorts E + H and E + G)
Description: Cmax of obinutuzumab was estimated from serum concentration data using non-compartmental analysis.
Time Frame: as for outcome 24
Population: Analysis was performed on all participants who received obinutuzumab (Cohort E+H and E+G) with measurable PK concentrations. Here, 'Overall Number of Participants Analyzed' signifies the number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Cohort E + Cohort H (DLBCL): Obinutuzumab + Polatuzumab | Cohort E + Cohort G (FL): Obinutuzumab + Polatuzumab
Number analyzed (Participants) | 40 | 35
mcg/mL | 340 (95.0) | 330 (87.9)

49. Secondary Outcome: Overall Survival (OS): Obinutuzumab-Containing Cohorts (Cohorts E + H and E + G)
Description: as for outcome 10
Time Frame: Baseline up to death due to any cause (from baseline up to study completion date, up to approximately 5.5 years)
Population: as for outcome 14
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort E + Cohort H (DLBCL): Obinutuzumab + Polatuzumab | Cohort E + Cohort G (FL): Obinutuzumab + Polatuzumab
Number analyzed (Participants) | 35 | 9
Months | 10.5 [5.5 to 16.7] | NA [38.4 to NA] — Median and corresponding CI could not be estimated because very few participants (<50%) had the event of interest.

50. Secondary Outcome: Percentage of Participants Who Died Due to Any Cause: Obinutuzumab Containing Cohorts (Cohorts E + H and E + G)
Description: Percentage of participants who died due to any cause was reported.
Time Frame: Baseline up to death due to any cause (from baseline up to study completion date, up to approximately 5.5 years)
Population: Obinutuzumab-Containing Cohorts (Cohorts E + H and E + G): Analysis was performed on efficacy-evaluable population.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort E + Cohort H (DLBCL): Obinutuzumab + Polatuzumab | Cohort E + Cohort G (FL): Obinutuzumab + Polatuzumab
Number analyzed (Participants) | 45 | 44
percentage of participants | 77.8 | 20.5

51. Secondary Outcome: Progression-free Survival (PFS) as Determined by Modified Response and Progression Criteria for NHL: Obinutuzumab Containing Cohorts (Cohorts E + H and E + G)
Description: as for outcome 8
Time Frame: Baseline up to PD or death due to any cause, whichever occurred first (up to approximately 5.5 years)
Population: Obinutuzumab-Containing Cohorts (Cohorts E + H and E + G): Analysis was performed on efficacy-evaluable population.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort E + Cohort H (DLBCL): Obinutuzumab + Polatuzumab | Cohort E + Cohort G (FL): Obinutuzumab + Polatuzumab
Number analyzed (Participants) | 45 | 44
months | 2.7 [2.1 to 5.9] | 19.5 [10.9 to 38.4]

52. Secondary Outcome: Percentage of Participants With PD as Determined by Modified Response and Progression Criteria for NHL or Death Due to Any Cause: Obinutuzumab Containing Cohorts (Cohorts E + H and E + G)
Description: as for outcome 7
Time Frame: Baseline up to PD or death due to any cause, whichever occurs first (up to approximately 5.5 years)
Population: Obinutuzumab-Containing Cohorts (Cohorts E + H and E + G): Analysis was performed on efficacy-evaluable population.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort E + Cohort H (DLBCL): Obinutuzumab + Polatuzumab | Cohort E + Cohort G (FL): Obinutuzumab + Polatuzumab
Number analyzed (Participants) | 45 | 44
percentage of participants | 88.9 | 56.8

ADVERSE EVENTS:
Time Frame: Baseline up to 30 days after the last dose of study treatment (up to approximately 12 months for rituximab-containing regimens [Arms A and B, Cohort C] and 24 weeks for Cohorts E, G, and H)
Description: Analysis was performed on safety-evaluable population.
Arm/Group | Arm A (FL+DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab | Arm B (FL+DLBCL): RTX+Polatuzumab,Then RTX+Pinatuzumab | Cohort C (FL): RTX + Polatuzumab | Cohort E (FL+DLBCL): Obinutuzumab + Polatuzumab | Cohort G (Expansion, FL): Obinutuzumab + Polatuzumab | Cohort H (Expansion, DLBCL): Obinutuzumab + Polatuzumab
All-Cause Mortality (participants affected / at risk) | 35/63 | 33/59 | 6/20 | 4/9 | 8/40 | 32/40
Serious Adverse Events (participants affected / at risk) | 27/63 | 21/59 | 8/20 | 3/9 | 9/40 | 18/40
Other Adverse Events (participants affected / at risk) | 63/63 | 58/59 | 20/20 | 9/9 | 37/40 | 38/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (FL+DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab (N=63) | Arm B (FL+DLBCL): RTX+Polatuzumab,Then RTX+Pinatuzumab (N=59) | Cohort C (FL): RTX + Polatuzumab (N=20) | Cohort E (FL+DLBCL): Obinutuzumab + Polatuzumab (N=9) | Cohort G (Expansion, FL): Obinutuzumab + Polatuzumab (N=40) | Cohort H (Expansion, DLBCL): Obinutuzumab + Polatuzumab (N=40)
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 2 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Colonic fistula (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 0
Duodenal perforation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Fistula of small intestine (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1
Hernial eventration (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Axillary pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 2 | 1 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 2 | 1 | 1 | 0 | 0 | 0
Sudden death (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hepatocellular injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hepatomegaly (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Clostridial sepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Febrile infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 1 | 0 | 2 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0 | 2 | 2
Sepsis (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Viral diarrhoea (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 2 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Wound secretion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Cachexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ganglioneuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 2 | 0 | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Liver Disorder (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hepatic Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (FL+DLBCL): RTX+Pinatuzumab,Then RTX+Polatuzumab (N=63) | Arm B (FL+DLBCL): RTX+Polatuzumab,Then RTX+Pinatuzumab (N=59) | Cohort C (FL): RTX + Polatuzumab (N=20) | Cohort E (FL+DLBCL): Obinutuzumab + Polatuzumab (N=9) | Cohort G (Expansion, FL): Obinutuzumab + Polatuzumab (N=40) | Cohort H (Expansion, DLBCL): Obinutuzumab + Polatuzumab (N=40)
Anaemia (Blood and lymphatic system disorders) | 9 | 10 | 1 | 2 | 4 | 4
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 19 | 15 | 8 | 4 | 8 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 2 | 0 | 0 | 4 | 4
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 1 | 1 | 2
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 3 | 3 | 0 | 0 | 2 | 0
Ear discomfort (Ear and labyrinth disorders) | 0 | 1 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 1 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 1 | 1 | 0 | 2 | 0
Dry eye (Eye disorders) | 2 | 0 | 0 | 0 | 3 | 0
Eye pain (Eye disorders) | 1 | 0 | 1 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 6 | 2 | 2 | 0 | 2 | 1
Visual impairment (Eye disorders) | 1 | 1 | 0 | 0 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 3 | 1 | 0 | 1 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 2 | 0 | 0 | 3 | 4
Abdominal pain (Gastrointestinal disorders) | 11 | 11 | 2 | 0 | 4 | 3
Abdominal pain lower (Gastrointestinal disorders) | 2 | 1 | 1 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 4 | 2 | 0 | 5 | 4
Constipation (Gastrointestinal disorders) | 18 | 14 | 5 | 0 | 14 | 8
Diarrhoea (Gastrointestinal disorders) | 28 | 25 | 5 | 3 | 13 | 14
Dry mouth (Gastrointestinal disorders) | 5 | 5 | 1 | 0 | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 4 | 8 | 3 | 0 | 5 | 3
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0 | 2 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 0 | 2 | 0 | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 2 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 20 | 25 | 11 | 0 | 11 | 14
Toothache (Gastrointestinal disorders) | 0 | 2 | 2 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 11 | 13 | 3 | 0 | 8 | 5
Asthenia (General disorders) | 11 | 16 | 0 | 1 | 3 | 8
Chest pain (General disorders) | 4 | 6 | 2 | 0 | 0 | 1
Chills (General disorders) | 5 | 4 | 3 | 0 | 8 | 5
Fatigue (General disorders) | 32 | 34 | 13 | 5 | 18 | 9
Feeling hot (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gait disturbance (General disorders) | 1 | 3 | 1 | 0 | 2 | 2
Influenza like illness (General disorders) | 0 | 8 | 0 | 1 | 1 | 0
Malaise (General disorders) | 1 | 2 | 1 | 0 | 2 | 1
Nodule (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 6 | 8 | 3 | 0 | 2 | 3
Pain (General disorders) | 5 | 1 | 3 | 0 | 0 | 1
Peripheral swelling (General disorders) | 1 | 2 | 0 | 0 | 2 | 0
Pyrexia (General disorders) | 15 | 9 | 5 | 2 | 5 | 3
Unevaluable event (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Seasonal allergy (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Candida infection (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 2
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 2
Infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 1 | 0 | 1 | 0
Mucosal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 2 | 2 | 1 | 0 | 0 | 2
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Pilonidal cyst (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 2 | 2 | 2 | 0
Tooth infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 5 | 2 | 3 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 6 | 2 | 0 | 0 | 3 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 0 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 2 | 0 | 0 | 3 | 2
Infusion related reaction (Injury, poisoning and procedural complications) | 3 | 1 | 2 | 1 | 7 | 3
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 2 | 0 | 1 | 3 | 1
Aspartate aminotransferase increased (Investigations) | 2 | 1 | 0 | 0 | 4 | 2
Blood creatinine increased (Investigations) | 2 | 1 | 0 | 1 | 1 | 1
Blood potassium decreased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 1
Neutrophil count decreased (Investigations) | 0 | 4 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 1 | 0 | 1 | 0 | 2
Protein total decreased (Investigations) | 0 | 0 | 0 | 0 | 2 | 0
Weight decreased (Investigations) | 6 | 7 | 3 | 1 | 0 | 0
Weight increased (Investigations) | 1 | 0 | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 1 | 4 | 0 | 1 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 13 | 17 | 4 | 0 | 7 | 5
Dehydration (Metabolism and nutrition disorders) | 6 | 3 | 2 | 0 | 4 | 2
Gout (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 2 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 4 | 2 | 1 | 1 | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 3 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 8 | 0 | 0 | 0 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 5 | 6 | 1 | 1 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 2 | 1 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 3 | 1 | 0 | 2 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 11 | 5 | 1 | 4 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 8 | 3 | 0 | 2 | 5
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 6 | 1 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Joint stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 6 | 2 | 0 | 3 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 6 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 2 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 6 | 3 | 0 | 2 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 12 | 4 | 1 | 7 | 6
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cluster headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Cubital tunnel syndrome (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 7 | 10 | 3 | 0 | 6 | 4
Dysgeusia (Nervous system disorders) | 2 | 3 | 1 | 0 | 3 | 0
Headache (Nervous system disorders) | 10 | 8 | 6 | 1 | 10 | 6
Hypoaesthesia (Nervous system disorders) | 3 | 2 | 2 | 0 | 1 | 1
Memory impairment (Nervous system disorders) | 1 | 3 | 2 | 0 | 0 | 0
Nerve compression (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 23 | 27 | 6 | 1 | 8 | 8
Paraesthesia (Nervous system disorders) | 5 | 1 | 2 | 0 | 4 | 3
Peripheral motor neuropathy (Nervous system disorders) | 2 | 5 | 1 | 0 | 4 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 16 | 17 | 11 | 2 | 7 | 2
Restless legs syndrome (Nervous system disorders) | 3 | 1 | 0 | 0 | 3 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 1 | 0 | 2 | 1
Adjustment disorder with depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 5 | 1 | 0 | 2 | 1
Depression (Psychiatric disorders) | 3 | 4 | 1 | 0 | 1 | 1
Hallucination olfactory (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 15 | 8 | 3 | 1 | 1 | 6
Dysuria (Renal and urinary disorders) | 1 | 3 | 1 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 15 | 3 | 1 | 7 | 6
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 0 | 2 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 11 | 11 | 2 | 0 | 5 | 8
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 2 | 0 | 1 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 2 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2 | 1 | 4 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 3 | 1 | 2 | 3
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 4 | 2 | 4 | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2 | 2 | 1 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 7 | 1 | 0 | 2 | 1
Brow ptosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0 | 0 | 0 | 3 | 2
Erythema (Skin and subcutaneous tissue disorders) | 4 | 1 | 1 | 0 | 3 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 4 | 0 | 0 | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 6 | 4 | 3 | 0 | 6 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 6 | 2 | 0 | 7 | 3
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 1 | 0
Thrombolysis (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 4 | 1
Haematoma (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 3 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 4 | 1 | 1 | 0 | 2 | 4
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 3 | 0 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 2 | 1 | 4 | 0 | 0 | 0
Skin Abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 1 | 0
Hepatic Encephalopathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Taste Disorder (Nervous system disorders) | 0 | 3 | 0 | 0 | 1 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-03): https://cdn.clinicaltrials.gov/large-docs/98/NCT01691898/Prot_SAP_000.pdf